CLINICAL TRIAL: NCT05336630
Title: SOCCER: Study Of forCeps Cannulation During ERcp
Brief Title: Study of Forceps Cannulation During ERCP
Acronym: SOCCER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Timothy Gardner, Principal Investigator, Staff Physician, Gastroenterology & Hepatology, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY02001449
Record Dates: First submitted 2022-04-14; First posted 2022-04-20 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Post-ERCP Acute Pancreatitis
MeSH Terms: interventions — Surgical Instruments

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either ERCP with forceps assisted cannulation or ERCP with no forceps.
Who Masked: Participant
Masking Description: Patients will be unblinded to their treatment on the 5 (+/- 2) day follow-up call.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Forceps Assisted Cannulation (Experimental): Patients will have a forceps assisted cannulation during their ERCPs.
  Interventions: Device: Forceps
- No Forceps Assisted Cannulation (No Intervention): Patients will not have a forceps assisted cannulation during their ERCPs.

INTERVENTIONS:
Device: Forceps — The forceps clears the redundant tissue to enable access to the papilla, as well as stabilizes the ampullary position to permit an easier cannulation. The forceps is an FDA approved instrument and does not put the patient at any higher risk for any adverse event. Please note that for the explicit purpose of the study the forceps will be used to grab tissue and not take biopsies. The forceps may still be used to take biopsies if the physician believes it is indicated.
  Arms: Forceps Assisted Cannulation

SUMMARY:
A difficult cannulation has been identified as one of the high risk factors for developing post-ERCP pancreatitis (PEP). The accessibility and morphology of the papilla influence the level of cannulation difficulty. The use of a forceps to assist in the cannulation is a demonstrated effective technique for cannulating papillae that are difficult to access. Thus, the objective of our study is to determine whether a forceps assisted cannulation leads to less difficult cannulation during ERCP. Because difficult cannulation is associated with increased risk of PEP, our study investigates whether the forceps assisted cannulation also reduces the incidence of PEP as a secondary outcome. Eligible patients who have consented will either be randomized to cannulation with forceps or cannulation with no forceps.

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP), an invasive procedure that combines endoscopy and x-ray to treat issues with the bile and pancreatic ducts, carries a two to ten percent risk of causing post-ERCP pancreatitis (PEP) [1]. Because acute pancreatitis is a devastating inflammatory condition that leads to extensive morbidity and mortality, efforts to reduce the risk of PEP in patients undergoing ERCP would enhance patient outcomes and would decrease the economic burden in treating PEP nationwide [2-4].

A difficult cannulation has been identified as one of the high risk factors for developing PEP [5]. A study performed by Scandinavian Association for Digestive Endoscopy (SADE) determined that cannulations with five or more attempts, a duration of five minutes or longer, or two or more unintended pancreatic duct (PD) wire passages significantly increased one's risk for PEP [6]. Thus, SADE defined a difficult cannulation as any cannulation with at least one of the following conditions: five or more attempts, five or more minutes, or two or more unintended PD wire passages [6]. This classification of a difficult cannulation has been adopted and standardized by the European Society of Gastrointestinal Endoscopy [7]. Because no current guidelines defining a difficult cannulation exist from the American College of Gastroenterology or American Gastroenterological Association, the European Society of Gastrointestinal Endoscopy (ESGE) guidelines as gathered from the SADE study are the worldwide standardized definition of difficult cannulation.

Difficult cannulations have been reported to occur at a frequency of 42 percent for all ERCP exams [8]. The morphology and accessibility of the papilla influence the level of difficulty. Some studies have indicated that different macroscopic appearances of the papilla result in varying cannulation difficulty levels. Based on a study gauging intraobserver and interobserver agreement to the macroscopic appearance of different papillae, papillae are categorized as: Type 1, normal appearing; Type 2, small; Type 3, protruding or pendulous; and Type 4, ridged or creased [9]. Haraldsson et al. found that Type 2 and Type 3 papillae were more difficult to cannulate [8]. Regardless of papilla type, the involvement of a trainee (a GI fellow) resulted in more difficult cannulations [8]. In addition, the presence of redundant tissue, such as periampullary diverticula-which occurs in up to 20 percent of patients undergoing ERCP-results in more challenging cannulations [10]. The use of a forceps to assist in the cannulation is a demonstrated effective technique for cannulating papillae that are difficult to access [10-12]. The forceps clears the redundant tissue to enable access to the papilla, as well as stabilizes the ampullary position to permit an easier cannulation [10]. Currently, no randomized controlled trials that detail to what extent a forceps facilitates cannulation exist. Thus, our study aims to determine whether a forceps assisted cannulation reduces the incidence of difficult cannulations and consequently PEP.

The primary outcome is difficult cannulation after randomization. A difficult cannulation will be defined as any cannulation that results in any of the following: 5 or more minutes, 5 or more cannulation attempts, or 2 or more unintentional pancreatic wire passages.

The secondary outcome is PEP. Acute pancreatitis according to the Atlanta guidelines, is at least two of the following: abdominal pain consistent with pancreatitis, lipase or amylase greater than 3 times the upper limit of normal, radiographic evidence of pancreatitis on cross sectional imaging [13].

The study intervention is the use of a forceps during the cannulation. Eligible patients who have consented will either be randomized to forceps assisted cannulation or no forceps used during cannulation. The forceps is an FDA approved instrument and does not put the patient at any higher risk for any adverse event.

SOCCER plans to enroll 152 patients. All patients undergoing ERCP at Dartmouth-Hitchcock endoscopy will be approached and consented for this study. Medical records will be reviewed to see if they meet inclusion/exclusion criteria. Patients will be consented day of the procedure. We received an approved HIPAA Authorization Waiver because access to a patient's chart will be required to determine inclusion/exclusion criteria.

Consent will be performed in the endoscopy pre-op area. During the standard of care ERCP, the patients will be randomized intraoperatively to either cannulation with forceps and cannulation with no forceps. Written informed consent will be reviewed and signed before any study related procedures are performed.

Please note that the primary outcome refers to a difficult cannulation AFTER randomization when the secondary inclusion criteria has been met. For example, if the secondary inclusion criteria met is difficult cannulation, then the primary outcome would be if from that point forward there were a difficult cannulation. As such, a total cannulation time of 10 minutes would enable the patient to be eligible (the first 5 minutes means the cannulation is difficult) and would mean the subject met the primary outcome (the second 5 minutes means cannulation after randomization is difficult). However, a total cannulation time of 8 minutes means the patient is eligible for the study (first 5 minutes means the cannulation is difficult) but did not meet the primary outcome (after randomization, the cannulation was not difficult because it was only 3 minutes). In a sense, the "difficult cannulation clock" is reset after randomization. If the secondary inclusion criteria met instead is papilla location or type, then the patient is randomized immediately before the cannulation and the difficult cannulation clock starts then. Measurement of difficult cannulation starts immediately after randomization upon the doctor's first cannulation attempt following randomization.

Randomization will occur in block format. Randomization assignments will be placed in sealed manila envelopes that will be opened at the time of randomization. Manila envelopes will be kept with the study coordinator.

After consent, data will be collected before, during, and after the procedure. The primary outcome will be measured during the procedure, whereas the secondary outcome will be determined during the 5 day follow up call. The study coordinator, GI fellow, or attending physician will call the patient 5 days (+/- 2 days) post-procedure to determine whether the patient developed PEP. Though it is preferred to contact the patient, other methods (chart review, emergency contact, outside records) are acceptable for determining the secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

PRIMARY INCLUSION CRITERIA:

* Patient consent
* ERCP done on native papilla

SECONDARY INCLUSION CRITERIA:

* Papilla in a diverticulum
* Papilla on rim of a diverticulum
* Difficult cannulation (5 attempts, 5 minutes, or 2 unintended PD wire passages)
* Redundant tissue overlying papilla
* Type 2, 3, or 4 papilla

Exclusion Criteria:

* Prior ampullectomy
* Known pregnancy, positive test, breastfeeding
* Clinical contraindication to ERCP
* Metal allergy
* Prior sphincterotomy
* Inability to follow protocol
* <18 years old
* Enrolled in another ERCP study
* Biliary/PD stent in place

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Gardner, MD MS, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Health, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thaker AM, Mosko JD, Berzin TM. Post-endoscopic retrograde cholangiopancreatography pancreatitis. Gastroenterol Rep (Oxf). 2015 Feb;3(1):32-40. doi: 10.1093/gastro/gou083. Epub 2014 Nov 17. PMID 25406464
- [Background] Neoptolemos JP, Raraty M, Finch M, Sutton R. Acute pancreatitis: the substantial human and financial costs. Gut. 1998 Jun;42(6):886-91. doi: 10.1136/gut.42.6.886. PMID 9691932
- [Background] Freeman ML, Nelson DB, Sherman S, Haber GB, Herman ME, Dorsher PJ, Moore JP, Fennerty MB, Ryan ME, Shaw MJ, Lande JD, Pheley AM. Complications of endoscopic biliary sphincterotomy. N Engl J Med. 1996 Sep 26;335(13):909-18. doi: 10.1056/NEJM199609263351301. PMID 8782497
- [Background] Elmunzer BJ, Serrano J, Chak A, Edmundowicz SA, Papachristou GI, Scheiman JM, Singh VK, Varadarajulu S, Vargo JJ, Willingham FF, Baron TH, Cote GA, Romagnuolo J, Wood-Williams A, Depue EK, Spitzer RL, Spino C, Foster LD, Durkalski V; SVI study group and the United States Cooperative for Outcomes Research in Endoscopy (USCORE). Correction to: Rectal indomethacin alone versus indomethacin and prophylactic pancreatic stent placement for preventing pancreatitis after ERCP: study protocol for a randomized controlled trial. Trials. 2020 Jun 3;21(1):471. doi: 10.1186/s13063-020-04458-0. PMID 32493506
- [Background] Freeman ML, Guda NM. Prevention of post-ERCP pancreatitis: a comprehensive review. Gastrointest Endosc. 2004 Jun;59(7):845-64. doi: 10.1016/s0016-5107(04)00353-0. No abstract available. PMID 15173799
- [Background] Halttunen J, Meisner S, Aabakken L, Arnelo U, Gronroos J, Hauge T, Kleveland PM, Nordblad Schmidt P, Saarela A, Swahn F, Toth E, Mustonen H, Lohr JM. Difficult cannulation as defined by a prospective study of the Scandinavian Association for Digestive Endoscopy (SADE) in 907 ERCPs. Scand J Gastroenterol. 2014 Jun;49(6):752-8. doi: 10.3109/00365521.2014.894120. Epub 2014 Mar 14. PMID 24628493
- [Background] Testoni PA, Mariani A, Aabakken L, Arvanitakis M, Bories E, Costamagna G, Deviere J, Dinis-Ribeiro M, Dumonceau JM, Giovannini M, Gyokeres T, Hafner M, Halttunen J, Hassan C, Lopes L, Papanikolaou IS, Tham TC, Tringali A, van Hooft J, Williams EJ. Papillary cannulation and sphincterotomy techniques at ERCP: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2016 Jul;48(7):657-83. doi: 10.1055/s-0042-108641. Epub 2016 Jun 14. PMID 27299638
- [Background] Haraldsson E, Kylanpaa L, Gronroos J, Saarela A, Toth E, Qvigstad G, Hult M, Lindstrom O, Laine S, Karjula H, Hauge T, Sadik R, Arnelo U. Macroscopic appearance of the major duodenal papilla influences bile duct cannulation: a prospective multicenter study by the Scandinavian Association for Digestive Endoscopy Study Group for ERCP. Gastrointest Endosc. 2019 Dec;90(6):957-963. doi: 10.1016/j.gie.2019.07.014. Epub 2019 Jul 18. PMID 31326385
- [Background] Haraldsson E, Lundell L, Swahn F, Enochsson L, Lohr JM, Arnelo U; Scandinavian Association for Digestive Endoscopy (SADE) Study Group of Endoscopic Retrograde Cholangio-Pancreaticography. Endoscopic classification of the papilla of Vater. Results of an inter- and intraobserver agreement study. United European Gastroenterol J. 2017 Jun;5(4):504-510. doi: 10.1177/2050640616674837. Epub 2016 Oct 17. PMID 28588881
- [Background] Levenick JM, Gardner TB, Hussain ZH, Gordon SR. SpyBite-assisted biliary cannulation for intradiverticular papilla during ERCP. Endoscopy. 2014;46 Suppl 1 UCTN:E514. doi: 10.1055/s-0034-1377365. Epub 2014 Nov 19. No abstract available. PMID 25409044
- [Background] Borahma M, Benelbarhdadi I, Berhili C, Lagdali N, Ajana FZ. Forceps-assisted technique: a new technique for difficult cannulation. Endoscopy. 2020 Jul;52(7):E247-E248. doi: 10.1055/a-1089-7418. Epub 2020 Jan 29. No abstract available. PMID 31995819
- [Background] Murabayashi T. The forceps-assisted technique for difficult cannulation has been in widespread use since 1996. Endoscopy. 2021 Apr;53(4):457. doi: 10.1055/a-1288-0801. Epub 2021 Mar 29. No abstract available. PMID 33780985
- [Background] Foster BR, Jensen KK, Bakis G, Shaaban AM, Coakley FV. Revised Atlanta Classification for Acute Pancreatitis: A Pictorial Essay. Radiographics. 2016 May-Jun;36(3):675-87. doi: 10.1148/rg.2016150097. PMID 27163588
- [Derived] Hadley SM Jr, Chevalier JI, Tomasetti GE, Hill JC, Duclos MC, Klibansky DA, Pohl H, Siegel CA, Toor A, Bensen SP, Adler JM, Gordon SR, Gardner TB. The Effectiveness of Forceps-Assisted Cannulation for Difficult Cannulation During Endoscopic Retrograde Cholangiopancreatography: Results of the SOCCER Randomized Controlled Trial. Am J Gastroenterol. 2026 Feb 1;121(2):337-344. doi: 10.14309/ajg.0000000000003531. Epub 2025 May 14. PMID 40367484

RESULTS

PARTICIPANT FLOW:
Groups:
- Forceps-assisted Group: Those who underwent cannulation with forceps-assisted technique
  n=70
  Age, years (SD) 61.9 (16.3)
  Gender Male, n (%) 33 (47.1) Female, n (%) 37 (52.9)
  BMI, kg/m2 29.3
  ERCP indication Choledocholithiasis, n (%) 29 (41.4) Extrahepatic malignant biliary obstruction, n (%) 20 (28.6) Intrahepatic malignant biliary obstruction, n (%) 4 (5.7) Chronic pancreatitis 2 (2.9) Sphincter of oddi dysfunction, n (%) 0 (0) Pancreatic stone disease, n (%) 0 (0) Bile leak, n (%) 5 (7.1) Pancreatic fistula, n (%) 1 (1.4) Dorsal duct intervention, n (%) 1 (1.4) Other, n (%) 8 (11.4)
  Trainee involvement, n (%) 43 (61.4)
  Papilla classification type I, n (%) 45 (64.3) II, n (%) 6 (8.6) III, n (%) 14 (20.0) IV, n (%) 5 (7.1)
  Papilla located within a diverticulum, n (%) 4 (5.7)
  Reason for randomization Failed initial cannulation, n (%) 35 (50.0) Papilla classification type, n (%) 21 (30.0) Papilla location, n (%) 14 (20.0)
- No Forceps-assisted Cannulation: Those who underwent cannulation without forceps-assisted technique
  n=81
  Age, years (SD) 68.3 (13.3)
  Gender Male, n (%) 32 (39.5) Female, n (%) 49 (60.5)
  BMI, kg/m2 27.5
  ERCP indication Choledocholithiasis, n (%) 37 (45.7) Extrahepatic malignant biliary obstruction, n (%) 19 (23.5) Intrahepatic malignant biliary obstruction, n (%) 4 (4.9) Chronic pancreatitis 2 (2.5) Sphincter of oddi dysfunction, n (%) 0 (0) Pancreatic stone disease, n (%) 0 (0) Bile leak, n (%) 4 (4.9) Pancreatic fistula, n (%) 1 (1.2) Dorsal duct intervention, n (%) 0 (0) Other, n (%) 14 (17.3)
  Trainee involvement, n (%) 51 (63.0)
  Papilla classification type I, n (%) 64 (79.0) II, n (%) 5 (6.2) III, n (%) 8 (9.9) IV, n (%) 4 (4.9)
  Papilla located within a diverticulum, n (%) 8 (9.9)
  Reason for randomization Failed initial cannulation, n (%) 45 (55.6) Papilla classification type, n (%) 11 (13.6) Papilla location, n (%) 25 (30.9)
Period: Overall Study
Arm/Group | Forceps-assisted Group | No Forceps-assisted Cannulation
Started | 70 (276 originally approached. 116 were screen fails, 8 declined consent, 72 did not meet difficult cannulation eligibility criteria and were thus excluded, 8 were excluded after consent for failure to reach eligibility criteria and 3 were excluded for miscellaneous reasons. 152 patients were therefore included in the study. Subsequently one patient was excluded due to inability to locate the papilla leaving 151 patients for final analysis) | 81 (276 originally approached. 116 were screen fails, 8 declined consent, 72 did not meet difficult cannulation eligibility criteria and were thus excluded, 8 were excluded after consent for failure to reach eligibility criteria and 3 were excluded for miscellaneous reasons. 152 patients were therefore included in the study. Subsequently one patient was excluded due to inability to locate the papilla leaving 151 patients for final analysis)
Completed | 70 (276 originally approached. 116 were screen fails, 8 declined consent, 72 did not meet difficult cannulation eligibility criteria and were thus excluded, 8 were excluded after consent for failure to reach eligibility criteria and 3 were excluded for miscellaneous reasons. 152 patients were therefore included in the study. Subsequently one patient was excluded due to inability to locate the papilla leaving 151 patients for final analysis) | 81 (276 originally approached. 116 were screen fails, 8 declined consent, 72 did not meet difficult cannulation eligibility criteria and were thus excluded, 8 were excluded after consent for failure to reach eligibility criteria and 3 were excluded for miscellaneous reasons. 152 patients were therefore included in the study. Subsequently one patient was excluded due to inability to locate the papilla leaving 151 patients for final analysis)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Same as assignment in participant flow
Groups:
- Forceps-assisted Group: n=70
  Age, years (SD) 61.9 (16.3)
  Gender Male, n (%) 33 (47.1) Female, n (%) 37 (52.9)
  BMI, kg/m2 29.3
  ERCP indication Choledocholithiasis, n (%) 29 (41.4) Extrahepatic malignant biliary obstruction, n (%) 20 (28.6) Intrahepatic malignant biliary obstruction, n (%) 4 (5.7) Chronic pancreatitis 2 (2.9) Sphincter of oddi dysfunction, n (%) 0 (0) Pancreatic stone disease, n (%) 0 (0) Bile leak, n (%) 5 (7.1) Pancreatic fistula, n (%) 1 (1.4) Dorsal duct intervention, n (%) 1 (1.4) Other, n (%) 8 (11.4)
  Trainee involvement, n (%) 43 (61.4)
  Papilla classification type I, n (%) 45 (64.3) II, n (%) 6 (8.6) III, n (%) 14 (20.0) IV, n (%) 5 (7.1)
  Papilla located within a diverticulum, n (%) 4 (5.7)
  Reason for randomization Failed initial cannulation, n (%) 35 (50.0) Papilla classification type, n (%) 21 (30.0) Papilla location, n (%) 14 (20.0)
- No Forceps-assisted Cannulation: n=81
  Age, years (SD) 68.3 (13.3)
  Gender Male, n (%) 32 (39.5) Female, n (%) 49 (60.5)
  BMI, kg/m2 27.5
  ERCP indication Choledocholithiasis, n (%) 37 (45.7) Extrahepatic malignant biliary obstruction, n (%) 19 (23.5) Intrahepatic malignant biliary obstruction, n (%) 4 (4.9) Chronic pancreatitis 2 (2.5) Sphincter of oddi dysfunction, n (%) 0 (0) Pancreatic stone disease, n (%) 0 (0) Bile leak, n (%) 4 (4.9) Pancreatic fistula, n (%) 1 (1.2) Dorsal duct intervention, n (%) 0 (0) Other, n (%) 14 (17.3)
  Trainee involvement, n (%) 51 (63.0)
  Papilla classification type I, n (%) 64 (79.0) II, n (%) 5 (6.2) III, n (%) 8 (9.9) IV, n (%) 4 (4.9)
  Papilla located within a diverticulum, n (%) 8 (9.9)
  Reason for randomization Failed initial cannulation, n (%) 45 (55.6) Papilla classification type, n (%) 11 (13.6) Papilla location, n (%) 25 (30.9)
- Total: Total of all reporting groups
Arm/Group | Forceps-assisted Group | No Forceps-assisted Cannulation | Total
Number analyzed (Participants) | 70 | 81 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (16.3) | 68.3 (13.3) | 65.0 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 32 | 69
  Male | 33 | 49 | 82
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — All patients were enrolled at Dartmouth-Hitchcock Medical Center in Lebanon, NH
  participants
    United States | 70 | 81 | 151
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.3 (7.4) | 27.5 (7.1) | 28.4 (7.2)
ERCP indication [Count of Participants; unit: Participants]
  Choledocholithiasis | 29 | 37 | 66
  Extrahepatic malignant biliary obstruction | 20 | 19 | 39
  Intrahepatic malignant biliary obstruction | 4 | 4 | 8
  Chronic pancreatitis | 2 | 2 | 4
  Sphincter of oddi dysfunction | 0 | 0 | 0
  Pancreatic stone disease | 0 | 0 | 0
  Bile leak | 5 | 4 | 9
  Pancreatic fistula | 1 | 1 | 2
  Dorsal duct intervention | 1 | 0 | 1
  Other | 8 | 14 | 22
Fellow involvement in ERCP procedure [Count of Participants; unit: Participants] | 43 | 51 | 94
Papilla morphologic classification type [Count of Participants; unit: Participants] — The papilla classification type is the standard consensus definition of the morphologic classification of the papilla. (I) Regular. (II) Small. (III) Protruding. (IV) Creased/ridged.
  Participants
    I | 45 | 64 | 109
    II | 6 | 5 | 11
    III | 14 | 8 | 22
    IV | 5 | 4 | 9
Reason for randomization [Count of Participants; unit: Participants]
  Failed initial cannulation | 35 | 45 | 80
  Papilla classification type | 21 | 11 | 32
  Papilla location | 14 | 25 | 39
Papilla located within a diverticulum [Count of Participants; unit: Participants] | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Cannulation Success Rate and Difficult Cannulation Rate
Description: A difficult cannulation will be defined as any cannulation that results in any of the following: 5 or more minutes, 5 or more cannulation attempts, or 2 or more unintentional pancreatic wire passages.
Time Frame: Baseline (during the ERCP)
Measure: Count of Participants; unit: Participants
Groups:
- Forceps-assisted Group: Forceps used during cannulation
- No Forceps-assisted Cannulation: No forceps used during cannulation
Arm/Group | Forceps-assisted Group | No Forceps-assisted Cannulation
Number analyzed (Participants) | 70 | 81
Participants
  Successful cannulation | 70 | 68
  Unsuccessful cannulation | 0 | 13

2. Secondary Outcome: Number of Post-ERCP Pancreatitis (PEP)
Time Frame: 5 (+/- 2) days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | Forceps-assisted Group | No Forceps-assisted Cannulation
Number analyzed (Participants) | 70 | 81
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the 5 +/- 2 day follow-up call.
Description: Adverse events were collected via chart review and patient contact
Groups:
- Forceps-assisted Group: n=70
- No Forceps-assisted Cannulation: n=81
Arm/Group | Forceps-assisted Group | No Forceps-assisted Cannulation
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/81
Serious Adverse Events (participants affected / at risk) | 5/70 | 9/81
Other Adverse Events (participants affected / at risk) | 2/70 | 2/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Forceps-assisted Group (N=70) | No Forceps-assisted Cannulation (N=81)
PEP (Hepatobiliary disorders) | 4 (4) | 3 (3) — Post-ERCP pancreatitis
Cholangitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Bile duct perforation (Hepatobiliary disorders) | 0 (0) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enceophalopathy (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Forceps-assisted Group (N=70) | No Forceps-assisted Cannulation (N=81)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Allergic reaction (General disorders) | 1 (1) | 0 (0) — mild allergic reaction, rash

LIMITATIONS AND CAVEATS:
ERCP procedure and postprocedure decisions were at the discretion of the attending endoscopist based on clinically appropriate guidelines. Another potential limitation is that the study did not account for multiple unintended biliary wire cannulations when the intent was PD wire cannulation. The results may not be as generalizable to endoscopists who are not as skilled with and comfortable using the forceps through the endoscope.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT05336630/Prot_SAP_000.pdf